CLINICAL TRIAL: NCT04542629
Title: Comparative Study of Dietary and Immunological Management of Refractory Epilepsy in Children Attending Assiut Pediatric University Hospital
Brief Title: Comparative Study of Dietary and Immunological Management of Refractory Epilepsy in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nancy Alaa, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSDIMRE
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Rituximab; Diet, Ketogenic; Trace Elements; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RITUXIMAB (Experimental): rituximab INTRAVENOUS 750MG/m2 every 2 weeks for 2 doses
  Interventions: Drug: RiTUXimab Injection [Rituxan]
- KETOGENIC DIET (Active Comparator): The common element of these different approaches is variable reduction in the amount of carbohydrate with appropriate increase in fat.
  Diets that produce a state of ketosis are referred to as ''ketogenic"
  Interventions: Drug: RiTUXimab Injection [Rituxan]
- TRACE ELEMENTS (Active Comparator): . Essential trace elements that include zinc, copper, magnesium, and selenium
  Interventions: Drug: RiTUXimab Injection [Rituxan]
- CORTICOSTEROID (Active Comparator): corticosteroid pulse therapy 30 mg /kg /day for 5 days monthly for 6 month
  Interventions: Drug: RiTUXimab Injection [Rituxan]

INTERVENTIONS:
Drug: RiTUXimab Injection [Rituxan] — 375 MG/M2 /WEEK INFUSION
  Other Names: KETOGENIC DIET; TRACE ELEMENTS; CORTICOSTEROID INJECTION

SUMMARY:
1. Comparison of the efficacy of Rituximab and ketogenic diet in controlling refractory seizures versus the traditional lines as corticosteroid and trace elements.
2. Improving the management of children with refractory seizures

DETAILED DESCRIPTION:
1. Definition of refractory epilepsy

   A task force of the International League Against Epilepsy proposed that drug-resistant epilepsy be defined as failure of adequate trials of two tolerated and appropriately chosen and used antiseizure drug schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom (1)

   . This requires application of the intervention at adequate strength/dosage for a sufficient length of time (2)..Terms refractory" intractable", drug-resistant" pharmaco-resistant" have been used interchangeably in several documented literature in different time periods (3). The first antiseizure drug fails in 20 to 40 percent of children with epilepsy; lack of efficacy and side effects contribute to treatment failure (4)

   Epidemiology About 10-20 % children with epilepsy develop drug refractory epilepsy (5).In a systematic review of 35 observational studies that included over 13,000 patients with epilepsy and 3900 patients with drug resistant epilepsy( DRE), the pooled prevalence of (DRE) was 30 percent, and the pooled incidence proportion was 15 percent (6).

   Risk factors

   - A high number of seizures prior to diagnosis and treatment

   - Genetic or inherited syndromes, for both generalized and localization-related epilepsy, have a better prognosis than symptomatic/cryptogenic epilepsy in both pediatric and adult populations (7).
   * Localization-related epilepsy underlies more than half of the cases of DRE in children (8,9).
   * Other findings more variably associated with the risk of DRE include a presentation with status epilepticus , a longer duration of epilepsy , a family history of epilepsy , a history of febrile convulsions , abnormal ( ELECTROENCEPHALOGRAM ) EEG findings . An abnormal neurologic examination and/or developmental delays (10,11).
   * Some pediatric studies have found that seizure onset in later childhood or adolescence appears to be more likely to be associated with DRE than seizures with onset between the ages of 5 and 10 years (12).

   Causes (13,14 ) Epilepsy syndromes

   Infancy

   • Epilepsy of infancy with migrating focal seizures
   * West syndrome
   * Dravet syndrome
   * Doose syndrome

   Childhood
   * Lennox-Gastaut syndrome
   * Epileptic encephalopathy with continuous spike and wave during sleep

   Metabolic

   • Pyridoxine dependent epilepsy

   • Biotinidase biosynthesis deficiency

   • Organic acidemia

   • Urea cycle disorders

   • Non-ketotic hyperglycinemia
   * Aminoacidopathies
   * Mitochondrial disorders including Alpers syndrome
   * Hashimoto encephalopathy

   Structural Abnormality

   • Malformations: Neuronal migration defects and neural tube defects

   • Neurocutaneous syndromes

   ,

   Infectious/Inflammatory:

   ,

   • Hypoxic ischemic encephalopathy,

   • Rasmussen encephalitis
   * Stroke
   * Tumors
   * Mesial temporal sclerosis

   Autoimmune epilepsies

   : N-methyl-D-aspartate receptor(NMDAR),

   Connective tissue disorders

   • Systemic lupus erythematosus,

   • Wegener's granulomatosis
   * , sarcoidsosis,
   * celiac disease,
   * Crohn's disease,
   * Behcet's
   * Sjorgren's syndrome,

   EVALUATION

   A- History and presentation :

   The approach depends upon age of onset, accurate description: pre-ictal, ictal, postictal events, precipitating events, seizure types, evolution relation to fever, previous history of febrile seizures (simple/complex), associated non-epileptic events, intake of (ANTI EPILPTIC DRUGS )AEDs with dose, developmental history, sleep history, detailed birth and peri-/antenatal history etc.

   B-Clinical examination depends upon anthropometry, syndromic facial dysmorphism, neurocutaneous features and detailed neurological and systemic assessment

   C- Pseudo-refractoriness indicates a condition in which seizures persist because the condition has not been adequately treated. The most common causes of pseudo refractory epilepsy include

<!-- -->

1. Inappropriate diagnosis

   -Cardiogenic (arrhythmias) and vasovagal events (syncope)
   * Parasomnias
   * Movement disorders (paroxysmal dyskinesias, cataplexy)
   * Psychogenic nonepileptic seizure (PNES) can mimic epileptic seizures. , do not respond to antiseizure drug therapy.

   While not without limitations, video-EEG monitoring is the gold standard test for the diagnosis of PNES
2. Bad compliance ; Missed dose
3. Incorrect drug An incorrect diagnosis of seizure classification leading to incorrect drug choice It is not uncommon for diopathic generalized epilepsy syndromes to be unrecognized and inappropriately treated with antiseizure drugs that are more appropriate to localization-related epilepsy .
4. Inadequate dosage
5. Inadequate frequency
6. Enzyme induction, especially if more than one antiepilptic drug AED or other medication is used
7. Inadequate anticonvulsant therapy

D-Investigation for the patients include;

1-EEG Routine EEG is a must for the clinical diagnosis of epilepsy and associated syndrome.

For the majority of patients with epilepsy, routine EEG is sufficient to classify seizure type and to start treatment But for refractory epilepsy ( RE) and a doubtful seizure, video-EEG monitoring is the best diagnostic tool available. 2-Drug level monitor 3-Serum electrolyte, serum glucose 4-MRI brain ; High-resolution MRI helps in isolating the cause of focal epilepsies and to predict long-term outcome and spontaneous remission in patients. In some cases, follow-up MRI reveals an etiology for epilepsy (such as cerebral neoplasm, autoimmune encephalitis) that was not seen on the initial study and requires specific therapies in addition to antiseizure drugs . 5- Metabolic Work up Arterial blood gas (ABG ) Serum ammonia ,lactate Tandem mass screening 6-Genetic Testing as karyotyping , gene sequence ,-Fundus examination The presence of features like dysmorphism, growth retardation, intellectual disability and hypotonia may indicate an underlying genetic syndrome, 7-CSF culture, analysis • Lumbar puncture of infectious process 8-vascuilitis panel Complete blood cell count Erythrocyte sedimentation rate CRP ( C REACTIVE PROTEIN ) VWF Ag (VON WILLEBRAND FACTOR) C 3, 4 (COMPLEMENT 3, 4) Antinuclear AB (ANTIBODY) Antiphospholipid AB Antineutrophil cytoplasmic AB Anti-DNA AB 9-autoimmune encephalitis (Hashimotos ) antithyroid peroxidase AB, anti-TSH receptor AB Anti-NMDA-R AB Anti-MOG AB (if CNS demyelination) abdominal ultrasound and -MRI abdomen;To detect ovarian teratoma as in autoimmune encephalitis

F-Practice recommendations for AED trial:

1. Optimise the dose of each AED by increasing the dose incrementally. If the maximum dose is ineffective introduce a second AED while continuing on the first. If seizure control is achieved, consider tapering the first AED. The advice to "start low and go slow" is appropriate 2. If one or two AEDs are ineffective, rational polytherapy should be explored. 3. Consider using AEDs with different mechanisms of action 4. Avoid using an AED that may worsen or provoke seizures Carbamazepine (CBZ), Oxcarbazepine (OXC), Phenytoin (PHT), Vigabatrin (VGB) and Tiagabine (TGB) may worsen myoclonus and absence seizures

   * Gabapentin (GBP) and Lamotrigine (LTG) may worsen myoclonus (Benzodiazepines given intravenously may worsen tonic seizures but may be very useful in treating Lennox-Gastaut and does not contraindicate their use

   Background A-Immunotherapy

   Evidence that the immune system is involved in the pathogenesis of epilepsy particularly, medically refractory epilepsy, has given rise to the use of adjunctive immunotherapy to slow or change the epileptogenic process.
   * The presumed immune therapeutic mechanism (ACTH, corticosteroids, plasmapheresis human immunoglobulin G, rituximab, azathioprine, and cyclophosphamide) is the removal of various neuroimmunological mechanisms involved. However, new models suggest suppression of endogenous brain agent's proconvulsant (neuropeptides) There is limited data of these treatments outside of specific epileptic encephalopathies such as West syndrome, Rasmussen encephalitis, Landau Kleffner and specific antibody mediated encephalitis such as anti NMDA encephalitis a) Corticosteroids: Their immunological mechanisms are inhibition diapedesis and therefore infiltration of lymphocytes to the injured areas, attenuating production of inflammatory humoral mediators (IL-2) and inhibition of leukocyte function (helper T lymphocytes mainly) as well as endothelial cells.

   Dose:

   Methylprednisolone 30 mg /kg /day for 5 days up to 1 gm /day ,pulsed monthly for 6 months (15).

   b) Plasmapheresis: the activity of auto-Abs can be modulated by treatment with IVIGs and by plasma treatment, which consists of the mechanical removal of Abs (16)

   c) Human immunoglobulin G:

   . IgGIV inhibits activation of innate cells, suppression of the production of proinflammatory cytokines, and soluble factors as tumor necrosis factor and interleukins induced by this factor. In endothelial cells and macrophages, suggesting a mechanism antiepileptic Dose:400 mg.kg /day for 5 days

   D--Rituximab:

   Rituximab, a chimeric monoclonal antibody that binds to CD20, was the first monoclonal antibody to be approved for clinical use in the therapy of cancer. It is approved for use against indolent B-cell non-Hodgkin's lymphoma (NHL), although its use has expanded significantly beyond that indication to virtually any CD20-positive NHL, and more recently into other areas such as autoimmune disorders

   ) Rituximab targets CD20, a transmembrane protein present on virtually all B cells from the stage at which they become committed to B-cell development until it is downregulated when they differentiate into antibody-secreting plasma cells (17) Numerous review articles whose primary focus is the action of rituximab in the treatment of RA, systemic lupus erythematosus (SLE) and other autoimmune diseases were published in 2006. Although there is a clear consensus that substantial clinical benefits are associated with rituximab therapy, the exact mechanism(s) by which the B-cell depletion promoted by rituximab ameliorates autoimmune disease activity remains an area of active discussion.(18, 19) The most likely mechanisms have naturally centered on the pathogenic role of B cells in autoimmune disease: these include the potential of B cells to give rise to plasma cells that secrete autoantibodies as well as the ability of autoantigen-specific B cells to present antigens to autoreactive T cells, which leads to T-cell activation, cytokine release and inflammation. In certain cases the results of clinical trials have demonstrated moderate correlations between reduction of autoantibody levels and lessening of disease symptoms, which has emphasized the role of autoantibodies in disease pathology. In other studies such correlations have not been observed, which has led investigators to favor B cell-T cell interactions as the most important in the etiology of tissue injury in autoimmune diseases.

(20 ,21)

B-Dietary Therapy

1. ketogenic diet rationale; The common element of these different approaches is variable reduction in the amount of carbohydrate with appropriate increase in fat.

   Diets that produce a state of ketosis are referred to as ''ketogenic" When deprived of glucose through restriction of carbohydrate intake, the human body begins metabolizing fat.In doing so, ketone bodies (acetoacetate, acetone, and hydroxybutyrate) are produced . (22).

   KDT is associated with increased mitochondrial biogenesis, oxidative phosphorylation, enhanced gamma-aminobutyric acid (GABA) levels, reduced neuronal excitability and firing, and stabilized synaptic function (23)

   Indicated Dietary therapy has been reported as effective in the treatment of seizures associated with glucose transporter 1 deficiency, pyruvate dehydrogenase deficiency, infantile spasms, absence epilepsy, myoclonic atonic epilepsy (Doose syndrome), Dravet syndrome, tuberous sclerosis complex, mitochondrial disorders, Lennox-Gastaut syndrome, Sturge-Weber syndrome, and Rett syndrome (24) Results from the randomized control trial indicated that 38% of children had more than 50% reduction in seizure frequency, and 7% had more than 90% reduction in seizure frequency three months after starting classic ketogenic diet. Retrospective studies reported a higher rate of seizure control (25).

   Contraindications Absolute contraindications for the use of diet therapy include carnitine deficiency (primary), carnitine palmitoyltransferase (CPT) I OR II deficiency, carnitine translocase deficiency, β-oxidation defects, pyruvate carboxylase deficiency, and porphyria.
2. trace elements and antioxidants; The equilibrium of trace elements is essential for a healthy nervous system due to their key roles in activation of specific enzyme in many pathways of the central nervous system function metabolism

   * Essential trace elements that include zinc, copper, magnesium, and selenium might play a role in the pathogenesis of seizures because of their possible influence on synaptogenesis, their actions on ligand- and voltage-gated ion channels, their effects on membrane lipid peroxidation and turnover of some neurotransmitters, and their roles in immunity (26)

Antioxidative defense mechanisms are important pathways involving trace elements. The accumulation of free radicals may lead to seizures and increases the risk o f their recurrence, because oxidative stress produces peroxidated membrane lipids and damages the cells

. Glutathione peroxidase (GPx) and superoxide dismutase (SOD) are two major enzymes that are involved in antioxidative defense mechanisms.

Selenium (Se), zinc (Zn), and copper (Cu) are important trace elements that participate in the structure of these enzymes patients with intractable epilepsy had significantly decreased levels of serum Se and Zn in comparison to the controlled group(27)

ELIGIBILITY:
Inclusion Criteria:

* 1-Age 1 month up to 17 years 2-Both male and female 3-Epileptic patient on two tolerated and appropriately chosen and used antiepilptic drugs with no response

Exclusion Criteria:

* 1-Neonate 2-Epieptic patient on monotherapy 3-Conditions mimic epilepsy 4-Pseudo refractioness 5-Absolute contraindications for the use of diet therapy include carnitine deficiency (primary), carnitine palmitoyltransferase (CPT) I OR II deficiency, carnitine translocase deficiency, β-oxidation defects, pyruvate carboxylase deficiency, and porphyria 6-Contraindication for Rituximab:

  1. Hypersensitivity to any component, murine proteins. b. Heart failure c. Active infection

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-20 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
a-seizure frequency b-antiepileptic drugs c-compliance to treatment d-number of hospital admission | 1 YEAR
  number of attacks of fits during monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Emad eldeen Mahmoud Hammad, professor, Study Director — aAssiut University Children Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Beleza P. Refractory epilepsy: a clinically oriented review. Eur Neurol. 2009;62(2):65-71. doi: 10.1159/000222775. Epub 2009 Jun 12. PMID 19521080
- [Background] Aneja S, Jain P. Refractory epilepsy in children. Indian J Pediatr. 2014 Oct;81(10):1063-72. doi: 10.1007/s12098-014-1533-1. Epub 2014 Aug 9. PMID 25106842
- [Background] Dudley RW, Penney SJ, Buckley DJ. First-drug treatment failures in children newly diagnosed with epilepsy. Pediatr Neurol. 2009 Feb;40(2):71-7. doi: 10.1016/j.pediatrneurol.2008.09.021. PMID 19135617
- [Background] Kalilani L, Sun X, Pelgrims B, Noack-Rink M, Villanueva V. The epidemiology of drug-resistant epilepsy: A systematic review and meta-analysis. Epilepsia. 2018 Dec;59(12):2179-2193. doi: 10.1111/epi.14596. Epub 2018 Nov 13. PMID 30426482
- [Background] Berg AT, Kelly MM. Defining intractability: comparisons among published definitions. Epilepsia. 2006 Feb;47(2):431-6. doi: 10.1111/j.1528-1167.2006.00440.x. PMID 16499772
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Dlugos DJ, Sammel MD, Strom BL, Farrar JT. Response to first drug trial predicts outcome in childhood temporal lobe epilepsy. Neurology. 2001 Dec 26;57(12):2259-64. doi: 10.1212/wnl.57.12.2259. PMID 11756607
- [Background] Berg AT, Shinnar S, Levy SR, Testa FM, Smith-Rapaport S, Beckerman B. Early development of intractable epilepsy in children: a prospective study. Neurology. 2001 Jun 12;56(11):1445-52. doi: 10.1212/wnl.56.11.1445. PMID 11402099
- [Background] Dlugos DJ. The early identification of candidates for epilepsy surgery. Arch Neurol. 2001 Oct;58(10):1543-6. doi: 10.1001/archneur.58.10.1543. PMID 11594910
- [Background] Brodie MJ, Barry SJ, Bamagous GA, Norrie JD, Kwan P. Patterns of treatment response in newly diagnosed epilepsy. Neurology. 2012 May 15;78(20):1548-54. doi: 10.1212/WNL.0b013e3182563b19. Epub 2012 May 9. PMID 22573629
- [Background] Nikodijevic D, Baneva-Dolnenec N, Petrovska-Cvetkovska D, Caparoska D. Refractory Epilepsy-MRI, EEG and CT scan, a Correlative Clinical Study. Open Access Maced J Med Sci. 2016 Mar 15;4(1):98-101. doi: 10.3889/oamjms.2016.029. Epub 2016 Feb 16. PMID 27275339
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] Eisenberg R, Albert D. B-cell targeted therapies in rheumatoid arthritis and systemic lupus erythematosus. Nat Clin Pract Rheumatol. 2006 Jan;2(1):20-7. doi: 10.1038/ncprheum0042. PMID 16932648
- [Background] Sfikakis PP, Boletis JN, Tsokos GC. Rituximab anti-B-cell therapy in systemic lupus erythematosus: pointing to the future. Curr Opin Rheumatol. 2005 Sep;17(5):550-7. doi: 10.1097/01.bor.0000172798.26249.fc. PMID 16093832
- [Background] Edwards JC, Cambridge G. B-cell targeting in rheumatoid arthritis and other autoimmune diseases. Nat Rev Immunol. 2006 May;6(5):394-403. doi: 10.1038/nri1838. PMID 16622478
- [Background] Cervenka MC, Kossoff EH. Dietary treatment of intractable epilepsy. Continuum (Minneap Minn). 2013 Jun;19(3 Epilepsy):756-66. doi: 10.1212/01.CON.0000431396.23852.56. PMID 23739109
- [Background] Bough KJ, Rho JM. Anticonvulsant mechanisms of the ketogenic diet. Epilepsia. 2007 Jan;48(1):43-58. doi: 10.1111/j.1528-1167.2007.00915.x. PMID 17241207
- [Background] Kossoff EH, Zupec-Kania BA, Rho JM. Ketogenic diets: an update for child neurologists. J Child Neurol. 2009 Aug;24(8):979-88. doi: 10.1177/0883073809337162. Epub 2009 Jun 17. PMID 19535814
- [Background] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. The ketogenic diet for the treatment of childhood epilepsy: a randomised controlled trial. Lancet Neurol. 2008 Jun;7(6):500-6. doi: 10.1016/S1474-4422(08)70092-9. Epub 2008 May 2. PMID 18456557
- [Background] Yuen AW, Sander JW. Can magnesium supplementation reduce seizures in people with epilepsy? A hypothesis. Epilepsy Res. 2012 Jun;100(1-2):152-6. doi: 10.1016/j.eplepsyres.2012.02.004. Epub 2012 Mar 8. PMID 22406257
- [Background] Hayashi M. Oxidative stress in developmental brain disorders. Neuropathology. 2009 Feb;29(1):1-8. doi: 10.1111/j.1440-1789.2008.00888.x. PMID 19154320
- [Background] Kanner AM, Soto A, Gross-Kanner H. Prevalence and clinical characteristics of postictal psychiatric symptoms in partial epilepsy. Neurology. 2004 Mar 9;62(5):708-13. doi: 10.1212/01.wnl.0000113763.11862.26. PMID 15007118
- [Background] van Mierlo P, Carrette E, Hallez H, Raedt R, Meurs A, Vandenberghe S, Van Roost D, Boon P, Staelens S, Vonck K. Ictal-onset localization through connectivity analysis of intracranial EEG signals in patients with refractory epilepsy. Epilepsia. 2013 Aug;54(8):1409-18. doi: 10.1111/epi.12206. Epub 2013 May 3. PMID 23647147
- [Background] Salmenpera TM, Symms MR, Rugg-Gunn FJ, Boulby PA, Free SL, Barker GJ, Yousry TA, Duncan JS. Evaluation of quantitative magnetic resonance imaging contrasts in MRI-negative refractory focal epilepsy. Epilepsia. 2007 Feb;48(2):229-37. doi: 10.1111/j.1528-1167.2007.00918.x. PMID 17295615